CLINICAL TRIAL: NCT04846231
Title: Supplements, Placebo, or Rosuvastatin Study
Acronym: SPORT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Version 1.0 23February2021
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hypercholesterolemia
Keywords: LDL & HDL Cholesterol, Statin, Dietary Supplements
MeSH Terms: conditions — Hypercholesterolemia | interventions — Fish Oils; Curcumin; Phytosterols; red yeast rice; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized 1:1:1:1:1:1:1:1 to the study groups in a blinded fashion. There will be 25 subjects per study group. The total sample size will be 200 patients.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects, investigator staff, persons performing the assessments, and the clinical trial team will be blinded to assigned study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Rosuvastatin (Active Comparator): 5 mg once per day
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): comparable to rosuvastatin 5 mg once per day
  Interventions: Other: Placebo
- Fish Oil (Active Comparator): Nature Made 2 soft gels per day
  Interventions: Dietary Supplement: Fish Oil, Cinnamon, Garlique,Turmeric, Plant Sterol, Red Yeast Rice
- Cinnamon (Active Comparator): 1200mg, 2 capsules per day
  Interventions: Dietary Supplement: Fish Oil, Cinnamon, Garlique,Turmeric, Plant Sterol, Red Yeast Rice
- Garlique (Active Comparator): Manufactured by Focus Consumer Health Marketgate,1 tablet per day
  Interventions: Dietary Supplement: Fish Oil, Cinnamon, Garlique,Turmeric, Plant Sterol, Red Yeast Rice
- Turmeric (Active Comparator): Bio Schwartz Turmeric Curcumin 1500 mg, 3 capsules per day
  Interventions: Dietary Supplement: Fish Oil, Cinnamon, Garlique,Turmeric, Plant Sterol, Red Yeast Rice
- Plant Sterol (Active Comparator): Nature Made CholestOff Plus, 2 soft gels twice a day
  Interventions: Dietary Supplement: Fish Oil, Cinnamon, Garlique,Turmeric, Plant Sterol, Red Yeast Rice
- Red Yeast Rice (Active Comparator): Arazo Nutrition 1200 mg, 2 capsules per day
  Interventions: Dietary Supplement: Fish Oil, Cinnamon, Garlique,Turmeric, Plant Sterol, Red Yeast Rice

INTERVENTIONS:
Dietary Supplement: Fish Oil, Cinnamon, Garlique,Turmeric, Plant Sterol, Red Yeast Rice — Subjects will be randomized to a Statin (Rosuvastatin 5 mg), a placebo, or a dietary supplement (Fish oil, Cinnamon, Garlic, Turmeric, Plant sterol, Red yeast rice).
  Arms: Cinnamon; Fish Oil; Garlique; Plant Sterol; Red Yeast Rice; Turmeric
Drug: Rosuvastatin — Subjects will be randomized to a Statin (Rosuvastatin 5 mg), a placebo, or a dietary supplement (Fish oil, Cinnamon, Garlic, Turmeric, Plant sterol, Red yeast rice).
  Other Names: Crestor
  Arms: Rosuvastatin
Other: Placebo — Subjects will be randomized to a Statin (Rosuvastatin 5 mg), a placebo, or a dietary supplement (Fish oil, Cinnamon, Garlic, Turmeric, Plant sterol, Red yeast rice).
  Arms: Placebo

SUMMARY:
A research study that is evaluating a low dose of an FDA approved statin medication in comparison to several commercially available over the counter dietary supplements which are marketed for cholesterol health. The study is comparing their effect on LDL cholesterol. LDL-cholesterol is low-density cholesterol and is sometimes referred to as "bad" cholesterol. Participants must live in Ohio and have a documented elevated LDL cholesterol level between 70-189mg/dL, must not currently be taking a statin or one of the dietary supplements included in the trial. Participants willing to discontinue a prohibited supplement for 4 weeks prior to enrollment will be allowed to participate. Trial participation is 4 weeks. Study medication will be provided at no charge. There will be 2 visits which include a lab draw at any Cleveland Clinic laboratory. Participants will be randomized (like a coin flip) to be in one of 8 possible groups: Rosuvastatin, Fish oil, Cinnamon, Garlic, Turmeric, Plant sterol, Red yeast rice, or placebo. The study will enroll 200 participants.

DETAILED DESCRIPTION:
Few well-controlled trials have studied the LDL-lowering effects of dozens of marketed "cholesterol health" dietary supplements. Prior research suggests most U.S. consumers believe cholesterol health supplements are safer than statins, and a majority of the public also believe supplements are as effective, or more effective, than prescription statins. Approximately one third of US adults who have been told they have elevated cholesterol are using a supplement to provide heart health protection rather than a statin. This represents a significant public health concern.

The purpose of this study is to evaluate the effect of select dietary supplements on cholesterol health compared with a low dose of a statin.

The study is comparing their effect on LDL and HDL cholesterol and inflammatory markers.

A randomized, single blind study design will be used to evaluate rosuvastatin 5 mg. vs. placebo and 6 commercially available over the counter supplements in a hierarchical testing order. Each participant will take study medication/supplement for a total of 4 weeks.

The study will randomize primary prevention patients who are considered borderline and intermediate risk for ASCVD based upon the 2018 Cholesterol Treatment Guidelines7 and are not taking any of the studied medication/supplements at the time of randomization.

Participants must have a documented elevated LDL cholesterol level between 70-189mg/dL, must not currently be taking a statin or one of the dietary supplements included in the trial. Participants willing to discontinue a prohibited supplement for 4 weeks prior to enrollment will be allowed to participate. Study medication will be provided at no charge. There will be 2 visits which include a lab draw at any Cleveland Clinic laboratory. Participants will be randomized (like a coin flip) to be in one of 8 possible groups: Rosuvastatin, Fish oil, Cinnamon, Garlic, Turmeric, Plant sterol, Red yeast rice, or placebo. The study will enroll 200 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. U.S. adults with primary hypercholesterolemia, 40-75 years of age.
3. Not currently taking statins or one of the dietary supplements included in the trial. Patients willing to discontinue a prohibited supplement for 4 weeks prior to enrollment will be allowed to participate.
4. LDL-cholesterol between 70 and 189 mg/dL.
5. Patients without diabetes mellitus and a 10-year risk of ASCVD between 5 and <20% using the pooled cohort risk equation. * Or Patients with diabetes mellitus in females 50-60 years of age or males 40-50 years of age with an LDL-C between 70-189 mg/dL and with an ASCVD risk below 20%.

Exclusion Criteria:

1. Age < 40 or >75 years of age
2. Women who are pregnant, plan to become pregnant within the next 6 months, or are breastfeeding.
3. Documented liver dysfunction or history of elevated LFTs indicating active liver disease
4. Documented chronic renal dysfunction within the past two years defined as an eGFR<30mL/min/m2.
5. Known hypersensitivity to rosuvastatin or any supplement under investigation (i.e. shellfish allergy, etc.).
6. Currently taking any prescription statin, or other prescription medication/supplements to treat elevated cholesterol or triglycerides.
7. Currently taking a medication/supplement that has known interaction with rosuvastatin, including fenofibrate, gemfibrozil, HIV medications, colchicine, cyclosporine, warfarin, anti-viral medications to treat Hepatitis C, regorafenib, and darolutamide.
8. Are unwilling to discontinue prohibited dietary supplement(s) for 4 weeks prior to participation or during the course of the trial. Other non-prohibited supplements will be permitted if doses have been stable for at least 4 weeks.
9. Known cardiovascular disease including a history of prior MI, stroke/TIA, PAD or prior revascularization procedures of the heart or vasculature (e.g. CABG, stenting, PCI etc.).
10. Fasting Triglycerides >200mg/dl.
11. In the opinion of the investigator, any other condition that will preclude participation in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luke Laffin, M.D., Principal Investigator — The Cleveland Clinic; Steven Nissen, M.D., Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laffin LJ, Bruemmer D, Garcia M, Brennan DM, McErlean E, Jacoby DS, Michos ED, Ridker PM, Wang TY, Watson KE, Hutchinson HG, Nissen SE. Comparative Effects of Low-Dose Rosuvastatin, Placebo, and Dietary Supplements on Lipids and Inflammatory Biomarkers. J Am Coll Cardiol. 2023 Jan 3;81(1):1-12. doi: 10.1016/j.jacc.2022.10.013. Epub 2022 Nov 6. PMID 36351465

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 203 subjects were enrolled and 199 randomized.
Period: Overall Study
Arm/Group | Rosuvastatin | Placebo | Fish Oil | Cinnamon | Garlique | Turmeric | Plant Sterol | Red Yeast Rice
Started | 25 | 25 | 24 | 25 | 25 | 25 | 25 | 25
Completed | 24 | 23 | 22 | 24 | 25 | 25 | 24 | 23
Not Completed | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin | Placebo | Fish Oil | Cinnamon | Garlique | Turmeric | Plant Sterol | Red Yeast Rice | Total
Number analyzed (Participants) | 25 | 25 | 24 | 25 | 25 | 25 | 25 | 25 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (6.02) | 63.5 (7.06) | 63.9 (6.48) | 65.7 (6.57) | 65.1 (4.93) | 65.1 (7.22) | 65.2 (5.30) | 64.2 (7.35) | 64.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 13 | 15 | 14 | 15 | 18 | 18 | 118
  Male | 11 | 14 | 11 | 10 | 11 | 10 | 7 | 7 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 25 | 25 | 24 | 25 | 25 | 24 | 25 | 25 | 198
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 2 | 0 | 2 | 2 | 4 | 18
  White | 22 | 22 | 20 | 23 | 24 | 22 | 23 | 21 | 177
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 24 | 25 | 25 | 25 | 25 | 25 | 199

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in LDL-C From Baseline for Rosuvastatin 5mg Daily Compared With Placebo and Each Dietary Supplement.
Description: The primary objective of this study is to compare the LDL lowering of rosuvastatin with the effect of six commonly used dietary supplements on cholesterol health.
Time Frame: The percent change in LDL-C for rosuvastatin 5 mg compared with dietary supplements after 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change LDL-C
Arm/Group | Rosuvastatin | Placebo | Fish Oil | Cinnamon | Garlique | Turmeric | Plant Sterol | Red Yeast Rice
Number analyzed (Participants) | 24 | 23 | 22 | 24 | 25 | 25 | 24 | 23
percent change LDL-C
  Percent change from baseline | -37.86 [-42.13 to -33.59] | -2.63 [-6.99 to 1.73] | -3.43 [-7.86 to 1.01] | 0.42 [-3.91 to 4.74] | 5.13 [0.97 to 9.29] | -1.29 [-5.44 to 2.87] | -4.37 [-8.65 to -0.09] | -6.55 [-10.94 to -2.16]
  Difference in Percent Change | 0 [0 to 0] | 35.22 [29.13 to 41.32] | 34.43 [28.28 to 40.58] | 38.27 [32.20 to 44.34] | 42.98 [37.02 to 48.95] | 36.57 [30.61 to 42.54] | 33.49 [27.42 to 39.55] | 31.31 [25.16 to 37.47]
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; To control the overall alpha of the study, the primary endpoint will be evaluated hierarchically. Each comparison to rosuvastatin will use an alpha of 0.05. This belongs to the primary endpoint; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 35.22, 95% CI 2-sided [29.13 to 41.32]
Statistical Analysis 2: Comparison: Rosuvastatin vs Fish Oil; To control the overall alpha of the study, the primary endpoint will be evaluated hierarchically. Each comparison to rosuvastatin will use an alpha of 0.05; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 34.43, 95% CI 2-sided [28.28 to 40.58]
Statistical Analysis 3: Comparison: Rosuvastatin vs Cinnamon; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 38.27, 95% CI 2-sided [32.20 to 44.34]
Statistical Analysis 4: Comparison: Rosuvastatin vs Garlique; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 42.98, 95% CI 2-sided [37.02 to 48.95]
Statistical Analysis 5: Comparison: Rosuvastatin vs Turmeric; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 36.57, 95% CI 2-sided [30.61 to 42.54]
Statistical Analysis 6: Comparison: Rosuvastatin vs Plant Sterol; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 33.49, 95% CI 2-sided [27.42 to 39.55]
Statistical Analysis 7: Comparison: Rosuvastatin vs Red Yeast Rice; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 31.31, 95% CI 2-sided [25.16 to 37.47]

2. Secondary Outcome: Percent Change in hsCRP for Rosuvastatin vs Dietary Supplements.
Description: Assess the effect of each supplement on inflammatory markers compared with rosuvastatin 5 mg.
Time Frame: The percent change in high sensitivity C reactive protein (hsCRP) for rosuvastatin 5 mg and dietary supplements compared with placebo after 4 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change hsCRP
Arm/Group | Rosuvastatin | Placebo | Fish Oil | Cinnamon | Garlique | Turmeric | Plant Sterol | Red Yeast Rice
Number analyzed (Participants) | 24 | 23 | 22 | 24 | 25 | 25 | 24 | 23
percent change hsCRP
  percentage change from baseline | -5.70 [-32.52 to 31.78] | -7.12 [-34.06 to 30.83] | -1.39 [-30.45 to 39.81] | 29.04 [-7.94 to 80.88] | 1.09 [-27.08 to 40.14] | -4.49 [-31.08 to 32.36] | -13.72 [-38.28 to 20.60] | 6.28 [-24.42 to 49.43]
  Difference in percent change | 0 [0 to 0] | -1.50 [-38.92 to 58.86] | 4.58 [-35.47 to 69.47] | 36.85 [-15.07 to 120.52] | 7.20 [-32.90 to 71.28] | 1.29 [-36.59 to 61.79] | -8.50 [-43.05 to 46.99] | 12.71 [-30.14 to 81.83]

3. Secondary Outcome: Percent Change in HDL-C, Total Cholesterol, and Triglycerides for Rosuvastatin vs Dietary Supplements.
Description: The percent change in HDL-C, total cholesterol, and triglycerides for each supplement compared with rosuvastatin.
  The percent change in HDL-C, total cholesterol, and triglycerides for each supplement compared with rosuvastatin. The percent change in HDL-C, total cholesterol, and triglycerides for each supplement compared with placebo.
Time Frame: After 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: % change HDLC,Tot Cholest, Triglycerides
Groups:
- Rosuvastatin: Rosuvastatin 5 mg once per day
- Placebo: Comparable to 5mg Rosuvastatin once per day
- Garlique: 1 tablet per day
- Turmeric: Bio Schwartz Curcumin, 1500mg, 3 capsules per day
- Plant Sterol: Nature Made CHolestOff Plus, 2 soft gels 2 times per day
- Red Yeast Rice: Arazo Nutrition, Red Yeast Rice, 1200mg, 2 capsules per day
Arm/Group | Rosuvastatin | Placebo | Fish Oil | Cinnamon | Garlique | Turmeric | Plant Sterol | Red Yeast Rice
Number analyzed (Participants) | 24 | 23 | 22 | 24 | 25 | 25 | 24 | 23
% change HDLC,Tot Cholest, Triglycerides
  Percent change from baseline HDL-C | 3.44 [-0.73 to 7.62] | 3.08 [-1.16 to 7.32] | 2.41 [-1.91 to 6.73] | -2.33 [-6.47 to 1.80] | 3.43 [-0.61 to 7.47] | 1.42 [-2.62 to 5.45] | -4.02 [-8.16 to 0.13] | 2.45 [-1.79 to 6.69]
  Difference in percentage change HDL-C | 0 [0 to 0] | -0.37 [-6.34 to 5.60] | -1.03 [-7.07 to 5.01] | -5.78 [-11.71 to 0.16] | -0.02 [-5.86 to 5.83] | -2.03 [-7.83 to 3.78] | -7.46 [-13.34 to -1.58] | -0.99 [-6.91 to 4.92]
  Percent change from baseline Total Cholesterol | -24.43 [-27.57 to -21.29] | -1.44 [-4.65 to 1.77] | -2.23 [-5.50 to 1.04] | 0.37 [-2.78 to 3.52] | 2.80 [-0.26 to 5.86] | -0.75 [-3.80 to 2.30] | -3.89 [-7.02 to -0.75] | -2.60 [-5.80 to 0.60]
  Difference in percent change Total Cholesterol | 0 [0 to 0] | 22.99 [18.49 to 27.48] | 22.20 [17.65 to 26.74] | 24.80 [20.36 to 29.23] | 27.23 [22.85 to 31.61] | 23.68 [19.30 to 28.06] | 20.54 [16.08 to 25.00] | 21.83 [17.33 to 26.33]
  Percent change from baseline Triglycerides | -19.25 [-27.60 to -9.94] | -1.41 [-11.78 to 10.18] | -5.01 [-15.19 to 6.40] | 8.34 [-2.80 to 20.75] | -5.43 [-15.03 to 5.26] | 0.26 [-9.82 to 11.47] | 1.28 [-9.17 to 12.93] | 4.11 [-6.81 to 16.31]
  Difference in percent change Triglycerides | 0 [0 to 0] | 22.09 [4.52 to 42.62] | 17.64 [0.58 to 37.58] | 34.16 [14.94 to 56.60] | 17.11 [0.41 to 36.60] | 24.16 [6.61 to 44.60] | 25.42 [7.49 to 46.35] | 28.93 [10.36 to 50.63]
Statistical Analysis 1: Comparison: Rosuvastatin; Test type: Superiority; p = 0.05, ANCOVA

4. Secondary Outcome: The Percent Change in HDL-C, Total Cholesterol, and Triglycerides for Placebo vs the Dietary Supplements.
Description: The percent change in HDL-C, total cholesterol, and triglycerides for each supplement compared with placebo.
Time Frame: After 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: % change HDLC, tot chole, triglycerides
Arm/Group | Rosuvastatin | Placebo | Fish Oil | Cinnamon | Garlique | Turmeric | Plant Sterol | Red Yeast Rice
Number analyzed (Participants) | 24 | 23 | 22 | 24 | 25 | 25 | 24 | 23
% change HDLC, tot chole, triglycerides
  Percent change from baseline HDL-C | 3.44 [-0.73 to 7.62] | 3.08 [-1.16 to 7.32] | 2.41 [-1.91 to 6.73] | -2.33 [-6.47 to 1.80] | 3.43 [-0.61 to 7.47] | 1.42 [-2.62 to 5.45] | -4.02 [-8.16 to 0.13] | 2.45 [-1.79 to 6.69]
  Difference in percent change HDL-C | 0.37 [-5.60 to 6.34] | 0 [0 to 0] | -0.67 [-6.68 to 5.35] | -5.41 [-11.31 to 0.49] | 0.35 [-5.49 to 6.19] | -1.66 [-7.52 to 4.20] | -7.09 [-13.07 to -1.12] | -0.63 [-6.67 to 5.42]
  Percent change from baseline total cholesterol | -24.43 [-27.57 to -21.29] | -1.44 [-4.65 to 1.77] | -2.23 [-5.50 to 1.04] | 0.37 [-2.78 to 3.52] | 2.80 [-0.26 to 5.86] | -0.75 [-3.80 to 2.30] | -3.89 [-7.02 to -0.75] | -2.60 [-5.80 to 0.60]
  Difference in percent change total cholesterol | -22.99 [-27.48 to -18.49] | 0 [0 to 0] | -0.79 [-5.34 to 3.76] | 1.81 [-2.71 to 6.33] | 4.24 [-0.19 to 8.68] | 0.69 [-3.75 to 5.13] | -2.45 [-6.95 to 2.06] | -1.16 [-5.69 to 3.37]
  Percent change from baseline triglycerides | -19.25 [-27.60 to -9.94] | -1.41 [-11.78 to 10.18] | -5.01 [-15.19 to 6.40] | 8.34 [-2.80 to 20.75] | -5.43 [-15.03 to 5.26] | 0.26 [-9.82 to 11.47] | 1.28 [-9.17 to 12.93] | 4.11 [-6.81 to 16.31]
  Difference in percent change triglycerides | -18.09 [-29.88 to -4.32] | 0 [0 to 0] | -3.65 [-17.77 to 12.90] | 9.88 [-5.92 to 28.34] | -4.08 [-17.78 to 11.91] | 1.69 [-12.79 to 18.58] | 2.73 [-12.16 to 20.14] | 5.60 [-9.79 to 23.63]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Rosuvastatin | Placebo | Fish Oil | Cinnamon | Garlique | Turmeric | Plant Sterol | Red Yeast Rice
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/24 | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25 | 1/24 | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 3/25 | 1/24 | 0/25 | 2/25 | 1/25 | 2/25 | 5/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=25) | Placebo (N=25) | Fish Oil (N=24) | Cinnamon (N=25) | Garlique (N=25) | Turmeric (N=25) | Plant Sterol (N=25) | Red Yeast Rice (N=25)
Clinical Change in Liver Function (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosuvastatin (N=25) | Placebo (N=25) | Fish Oil (N=24) | Cinnamon (N=25) | Garlique (N=25) | Turmeric (N=25) | Plant Sterol (N=25) | Red Yeast Rice (N=25)
Muscle Pain / Tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT04846231/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT04846231/SAP_001.pdf